CLINICAL TRIAL: NCT02923726
Title: Assessment of Primary Prevention Patients Receiving An ICD - Systematic Evaluation of ATP (APPRAISE ATP)
Brief Title: Assessment of Primary Prevention Patients Receiving An ICD - Systematic Evaluation of ATP
Acronym: APPRAISE ATP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C1924
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Sudden Cardiac Death
Keywords: Antitachycardia Pacing Therapy; Shock Therapy; Primary Prevention
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATP and Shock (Active Comparator): Once tachycardia has been detected and duration met, this group would receive antitachycardia pacing prior to shock therapy.
  Interventions: Device: Arm 1 (ATP+Shock)
- Shock only (Experimental): Once tachycardia has been detected and duration met, this group would receive shock therapy only.
  Interventions: Device: Arm 2 (shock only)

INTERVENTIONS:
Device: Arm 1 (ATP+Shock) — Subjects will be randomized and device programmed to the respective arm.
  Arms: ATP and Shock
Device: Arm 2 (shock only) — Subjects will be randomized and device programmed to the respective arm.
  Arms: Shock only

SUMMARY:
The primary objective is to understand the role of antitachycardia pacing (ATP) in primary prevention patients indicated for implantable cardioverter-defibrillator (ICD) therapy and programmed according to current guidance of higher rate cut-offs and therapy delays. The time to first all-cause shock will be tested in subjects with standard therapy (ATP and shocks) compared to subjects programmed to shock only to assess equivalency.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a Boston Scientific transvenous ICD (de novo implant or upgrade from pacemaker to ICD) implanted because of one of the following:

  * Prior myocardial infarction (MI) and left ventricular ejection fraction (LVEF) ≤ 30% OR
  * Ischemic or non-ischemic cardiomyopathy, and LVEF ≤ 35%, and a New York Heart Association (NYHA) class II or III
* Subject is age 21 or above, or is considered of legal age per given geography
* Subject is willing and capable of providing informed consent
* Subject is willing and capable of complying with follow-up visits as defined by this protocol

Exclusion Criteria:

* History of spontaneous sustained Ventricular Tachycardia (VT) (≥ 160 bpm at ≥ 30 seconds in duration) or Ventricular Fibrillation (VF) not due to a reversible cause
* NYHA Class IV documented in the medical records within 90 calendar days prior to enrollment
* Subject is eligible and scheduled for cardiac resynchronization (CRT) implant
* Subjects with a previous subcutaneous ICD (S-ICD)
* Subject with existing transvenous ICD (TV-ICD) device implanted for greater than 60 days
* Subjects with coronary artery bypass graft surgery or percutaneous coronary intervention within the past 90 calendar days prior to enrollment
* Subjects with documented myocardial infarction within the past 90 calendar days prior to enrollment
* Subjects on the active heart transplant list
* Subject who has a ventricular assist device (VAD) or is to receive a VAD
* Life expectancy shorter than 18 months due to any medical condition (e.g., cancer, uremia, liver failure, etc…)
* Subjects currently requiring hemodialysis
* Subject who is known to pregnant or plans to become pregnant over the course of the trial
* Subject is enrolled in any other concurrent clinical study, with the exception of local mandatory governmental registries and observational studies/registries, without the written approval from Boston Scientific

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2692 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Schuger, M.D., Principal Investigator — University of Rochester Clincal Cardiovascular Research Center
Locations (134):
- United States (89):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Tri-City Cardiology, Mesa, Arizona
  - Cardiovascular Consultants, LTD, Phoenix, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Mercy Clinic Cardiology, Rogers, Arkansas
  - Comprehensive Cardiovascular Specialists, Alhambra, California
  - Scripps Mercy Chula Vista, Chula Vista, California
  - VA Loma Linda, Loma Linda, California
  - Cardiovascular Consultants Medical Group, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Cardiac Specialists, Danbury, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Bradenton Cardiology, Bradenton, Florida
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - St Vincent's Medical Center, Jacksonville, Florida
  - Heart of the Villages, Lady Lake, Florida
  - Watson Clinic Center for Research, Inc, Lakeland, Florida
  - Charlotte Heart & Vascular, Port Charlotte, Florida
  - Brevard Cardiovascular Research Associates, Inc, Rockledge, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - AdventHeatlh Tampa, Tampa, Florida
  - CorVita Science Foundation, Chicago, Illinois
  - Adventist Hinsdale Hospital, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Lutheran Medical Group, Fort Wayne, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Hospital Medical Center, West Des Moines, Iowa
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Richard A. Henson Research Institute of Peninsula Regional Medical Center, Salisbury, Maryland
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - Southcoast Physicians Group, Fall River, Massachusetts
  - Mass Heart and Rhythm, Leominster, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Western Michigan University - Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Great Lakes Heart & Vascular Institute, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - St. Luke's Hospital of Duluth, Duluth, Minnesota
  - Heart and Vascular Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cox Health, Springfield, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardiovascular Associates of the Delaware Valley., Haddon Heights, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - St. Joseph's Region Medical Center, Paterson, New Jersey
  - Weill Cornell Medical University, New York, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Regional Cardiac Arrhythmia, Inc, Steubenville, Ohio
  - Mount Carmel Columbus Cardiology Consultants, Westerville, Ohio
  - Lehigh Valley Hospital Pocono, Allentown, Pennsylvania
  - Bryn Mawr Medical Specialists, Bryn Mawr, Pennsylvania
  - The Arrhythmia Institute, Newtown, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - McLeod Cardiology Associates, Florence, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota
  - VA North Texas Health Care System in Dallas, Dallas, Texas
  - Apex Trials Group, LLC, Fort Worth, Texas
  - University of Texas Houston Health Science Center, Houston, Texas
  - Heart Institute of East Texas, Lufkin, Texas
  - Mission Research Institute, New Braunfels, Texas
  - McKay Dee Cardiology, Ogden, Utah
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - VA Salt Lake City Health System, Salt Lake City, Utah
  - Bon Secours Heart & Vascular Institute, Mechanicsville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Cardiovascular Specialist, Richmond, Virginia
  - Providence Regional Medical Centre Everett, Everett, Washington
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Bellin Health, Green Bay, Wisconsin
- Austria (2):
  - Kepler Universitaetsklinikum GmbH, Linz
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Canada (8):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Scarborough Health Network-Centenary Site, Scarborough Village, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec., Québec, Quebec
- Italy (6):
  - Policlinico di Modena, Modena, Emilia-Romagna
  - Osp. Civile S. Maria Delle Grazie, Pozzuoli, Southern Cluster
  - Presidio Ospedale San Giovanni Bosco, Napoli
  - Hospital Buon Consiglio, Napoli
  - Ospedale dei Pellegrini, Napoli
  - Az. Osp. S. Andrea, Rome
- Japan (9):
  - Chiba University Hospital, Chiba, Chiba
  - Kokura Memorial Hospital, Kitakyushu-Shi, Fukuoka
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto-shi,
  - Tachikawa General Hospital, Nagaoka-shi, Niigata
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - National Crebral and Cardiovascular Center Hospital, Suita, Osaka
  - Saitama Medical University International Medical Cnter, Hidaka-shi, Saitama
- South Korea (12):
  - Chonnam National University, Gwangju, Donggu
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsang
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Donostia, San Sebastián
- United Kingdom (5):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Liverpool Heart and Chest - LHCH, Liverpool
  - St. Bartholomew's Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuger C, Joung B, Ando K, Mont L, Lambiase PD, O'Hara GE, Jennings JM, Yung D, Boriani G, Piccini JP, Wold N, Stein KM, Daubert JP; APPRAISE ATP Investigators. Assessment of Antitachycardia Pacing in Primary Prevention Patients: The APPRAISE ATP Randomized Clinical Trial. JAMA. 2024 Nov 26;332(20):1723-1731. doi: 10.1001/jama.2024.16531. PMID 39361311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for participants began on 30 Sep 2016 and ended on 13 Apr 2021 when the adjudicated primary episode target had been met. Potential participants, located at medical clinics or hospitals, were eligible for the study if they were 21 years of age or older and had a Class 1 or IIA indication for primary prevention implantable cardioverter defibrillator (ICD) therapy with a low left ventricular ejection fraction. Participants were considered enrolled once consented.
Pre-assignment Details: Of the 2692 participants enrolled,19 were consent ineligible and 12 were intent and therefore not randomized. 2595 participants were randomized.
  Consented and Ineligible: Consent signed but eligibility criteria was not met at time of enrollment
  • Intent: All eligibility criteria met and consent signed, but participant was not randomized due to:
  * no longer meeting eligibility criteria at the time of randomization
  * no longer willing to participate in the study
Period: Overall Study
Arm/Group | ATP and Shock | Shock Only
Started | 1302 | 1293
Completed | 769 | 811
Not Completed | 533 | 482
Not completed — Death | 196 | 175
Not completed — Withdrawal by Subject | 337 | 307

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATP and Shock | Shock Only | Total
Number analyzed (Participants) | 1302 | 1293 | 2595
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (11.5) | 63.8 (11.1) | 63.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data missing for one randomized subject in the ATP and Shock arm.
  Participants
    number analyzed (Participants) | 1301 | 1293 | 2594
    Female | 277 | 304 | 581
    Male | 1024 | 989 | 2013
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data was not reported for 26 subjects. The total number analyzed for both arms has been adjusted to remove these subjects.
  Participants
    Race: number analyzed (Participants) | 1287 | 1282 | 2569
    Race: American Indian or Alaksa Native | 5 | 8 | 13
    Race: Asian | 209 | 206 | 415
    Race: Black or African Heritage | 169 | 178 | 347
    Race: Caucasian | 860 | 849 | 1709
    Race: Hispanic or Latino | 39 | 37 | 76
    Race: Native Hawaiian or Pacific Islander | 2 | 3 | 5
    Race: Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants] — All data was available for region of enrollment, so the number analyzed is the total population for both arms. Population: Data was not reported for 17 subjects. The total number analyzed for both arms has been adjusted to remove these subjects.
  Participants
    Canada: number analyzed (Participants) | 1294 | 1284 | 2578
    Canada | 141 | 151 | 292
    Austria | 13 | 15 | 28
    South Korea | 123 | 129 | 252
    United States | 841 | 823 | 1664
    Japan | 65 | 60 | 125
    Italy | 71 | 71 | 142
    United Kingdom | 20 | 17 | 37
    Spain | 20 | 18 | 38
History of Atrial Fibrillation [Count of Participants; unit: Participants]
  Permanent Atrial Fibrillation | 70 | 56 | 126
  Persistent Atrial Fibrillation | 95 | 92 | 187
  Paroxysmal Atrial Fibrillation | 176 | 208 | 384
  No History of Atrial Fibrillation | 961 | 937 | 1898
Etiology [Count of Participants; unit: Participants]
  Ischemic | 757 | 753 | 1510
  Non-ischemic | 545 | 540 | 1085
Diabetes [Count of Participants; unit: Participants] | 525 | 520 | 1045
Device Type [Count of Participants; unit: Participants] — Population: Data was missing for one subject in the Shock Only arm and two subjects in the ATP +Shock arm.
  Participants
    number analyzed (Participants) | 1300 | 1292 | 2592
    Single Chamber ICD | 678 | 646 | 1324
    Dual Chamber ICD | 622 | 646 | 1268
Indication [Count of Participants; unit: Participants] — All data was available for indications in both arms so the number analyzed is the total population for both arms.
  Participants
    Myocardial Infarction (MI) and Ejection Fraction (EF) >/= 30% | 417 | 445 | 862
    New York Heart Association (NYHA) Class II/III and EF </= 35% | 876 | 842 | 1718
    Other | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Shock
Description: The incidence of all-cause shocks in subjects programmed with shocks only will be compared with subjects programmed to standard therapy (ATP and shock) to assess equivalency. All shocks delivered by the device were adjudicated by an external committee as to whether they were appropriately or inappropriately delivered. All shocks, appropriate and inappropriate, contributed to the evaluation of this endpoint.
Time Frame: 5 years
Population: All randomized subjects.
Measure: Count of Participants; unit: Participants
Groups:
- ATP and Shock: Receive antitachycardia pacing prior to shock therapy.
- Shock Only: Receive shock therapy only.
Arm/Group | ATP and Shock | Shock Only
Number analyzed (Participants) | 1302 | 1293
Participants | 129 | 178
Statistical Analysis 1: Comparison: ATP and Shock vs Shock Only; Test type: Superiority; p = 0.005, Log Rank; Hazard Ratio (HR) = 0.72, 95.9% CI 2-sided [0.57 to 0.92] — Shock only was the reference group. Confidence interval adjusted for interim analyses

2. Secondary Outcome: All-Cause Shock or Death From Any Cause
Description: incidence of all-cause shocks or death from any cause
Time Frame: 5 years
Population: All randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ATP and Shock | Shock Only
Number analyzed (Participants) | 1302 | 1293
Participants | 297 | 322
Statistical Analysis 1: Comparison: ATP and Shock vs Shock Only; Test type: Superiority; p = 0.284, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.78 to 1.07] — Shock Only was the reference group

3. Secondary Outcome: Appropriate Shock
Description: incidence of first appropriate shock All shocks delivered by the device were adjudicated by an external committee as to whether they were appropriately or inappropriately delivered. Appropriate shocks contributed to the evaluation of this endpoint.
Time Frame: 5 years
Population: Randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ATP and Shock | Shock Only
Number analyzed (Participants) | 1302 | 1293
Participants | 96 | 132
Statistical Analysis 1: Comparison: ATP and Shock vs Shock Only; Test type: Superiority; p = 0.020, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.56 to 0.95] — Shock Only arm is reference group

4. Secondary Outcome: Inappropriate Shock
Description: incidence of first inappropriate shock All shocks delivered by the device were adjudicated by an external committee as to whether they were appropriately or inappropriately delivered. Inappropriate shocks contributed to the evaluation of this endpoint.
Time Frame: 5 years
Population: All randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ATP and Shock | Shock Only
Number analyzed (Participants) | 1302 | 1293
Participants | 40 | 62
Statistical Analysis 1: Comparison: ATP and Shock vs Shock Only; Test type: Superiority; p = 0.033, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.44 to 0.97] — Shock Only is the reference group

5. Secondary Outcome: All Cause Mortality
Description: incidents of all cause mortality
Time Frame: 5 years
Population: All randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ATP and Shock | Shock Only
Number analyzed (Participants) | 1302 | 1293
Participants | 196 | 174
Statistical Analysis 1: Comparison: ATP and Shock vs Shock Only; Test type: Superiority; p = 0.184, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.94 to 1.41] — Shock Only is the reference group

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from time of enrollment through a common end date and a median follow-up time of 40 months.
Description: Adverse events and deaths occurring after 5 years of follow-up are included; therefore, there may be more events reported here than in the endpoints.
  Acronyms:
  RA: right atrial PG: pulse generator RV: right ventricle DFT: defibrillation threshold testing SVT: supraventricular tachycardia AVRT: atrioventricular reentrant tachycardia AVNRT: atrioventricular nodal reentrant tachycardia EAT: ectopic atrial tachycardia ERI: elective replacement indicator
Arm/Group | ATP and Shock | Shock Only
All-Cause Mortality (participants affected / at risk) | 196/1302 | 175/1293
Serious Adverse Events (participants affected / at risk) | 633/1302 | 618/1293
Other Adverse Events (participants affected / at risk) | 420/1302 | 448/1293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATP and Shock (N=1302) | Shock Only (N=1293)
Unable to capture - RA PG System (Product Issues) | 0 (0) | 1 (1)
Elevated threshold - RV PG System (Product Issues) | 0 (0) | 1 (1)
Impedance Out of Range - RV PG System (Product Issues) | 1 (1) | 0 (0)
Undersensing - Defibrillation - PG System (Product Issues) | 2 (2) | 0 (0)
Elevated DFT - Defibrillation - PG System (Product Issues) | 1 (1) | 0 (0)
Inappropriate Tachy Therapy - SVT - PG System Therapy (Product Issues) | 13 (14) | 17 (18)
Infection (>30 days post-implant) - PG System - Subject related (Infections and infestations) | 9 (9) | 7 (7)
Twiddler's Syndrome - PG System - Subject related (Psychiatric disorders) | 2 (2) | 0 (0)
Migration - PG System - Subject related (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post-surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-surgical infection (<=30 days post-implant) (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Chest pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Death-Unknown - PG System - Procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep Vein Thrombosis - PG System - Procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unable to capture - RA Lead (Product Issues) | 0 (0) | 1 (1)
Conductor coil fracture - RA Lead (Product Issues) | 1 (1) | 0 (0)
Myocardial perforation post-implant - RA Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - RA Lead (Product Issues) | 1 (1) | 0 (0)
Dislodgment - No reported signs - RA Lead (Product Issues) | 1 (1) | 0 (0)
Thrombosis - Lead (Product Issues) | 1 (1) | 0 (0)
Tricuspid Valve Damage RV lead - Lead (Product Issues) | 1 (1) | 0 (0)
Unable to capture - RV Lead (Product Issues) | 0 (0) | 1 (1)
Extracardiac stimulation - RV Lead (Product Issues) | 1 (1) | 0 (0)
Conductor coil fracture - RV Lead (Product Issues) | 1 (1) | 1 (1)
Myocardial perforation post-implant - RV Lead (Product Issues) | 2 (2) | 2 (2)
Dislodgment - Unable to capture - RV Lead (Product Issues) | 0 (0) | 2 (2)
Dislodgment - Elevated threshold -RV Lead (Product Issues) | 2 (2) | 3 (3)
Dislodgment - Oversensing - RV Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - RV Lead (Product Issues) | 1 (1) | 1 (1)
Dislodgment - No reported signs - RV Lead (Product Issues) | 2 (2) | 1 (1)
Impedance Out of Range - Defibrillation lead (Product Issues) | 0 (0) | 1 (1)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pericardial effusion - Procedure (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
3rd degree AV block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Pulseless Electrical Activity (PEA) (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (VF) (Cardiac disorders) | 24 (25) | 27 (30)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 43 (71) | 49 (57)
Nonsustained Ventricular Tachycardia (NSVT) (Cardiac disorders) | 3 (3) | 3 (3)
Atrial Fibrillation (AF) (Cardiac disorders) | 43 (57) | 68 (84)
Atrial Flutter (Cardiac disorders) | 8 (8) | 5 (5)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 5 (6) | 6 (7)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 4 (4) | 7 (8)
SVT vs VT - Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
VF with Syncope - Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
VT with Syncope - Arrhythmia (Cardiac disorders) | 9 (9) | 15 (15)
Syncope - Heart failure (Cardiac disorders) | 1 (1) | 2 (2)
Dizziness - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - Heart failure (Cardiac disorders) | 8 (8) | 5 (7)
Dyspnea - Heart failure (Cardiac disorders) | 34 (44) | 48 (58)
Peripheral edema - Heart failure (Cardiac disorders) | 2 (2) | 7 (7)
Pulmonary edema - Heart failure (Cardiac disorders) | 4 (4) | 4 (4)
Fatigue - Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Renal insufficiency/failure - Heart failure (Cardiac disorders) | 2 (2) | 4 (4)
Dehydration - Heart failure (Cardiac disorders) | 3 (3) | 0 (0)
Gastrointestinal - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension - Heart failure (Cardiac disorders) | 1 (1) | 3 (3)
Pleural Effusion - Heart failure (Cardiac disorders) | 1 (1) | 7 (8)
Cardiac medication complication - Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 46 (55) | 56 (65)
Multiple heart failure symptoms (Cardiac disorders) | 171 (248) | 160 (285)
Hypertension - Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Heart transplant - Heart Failure Patient Condition - Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Multi-system failure - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 13 (14) | 12 (13)
Hypertension/Hypertensive Crisis (Vascular disorders) | 5 (5) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 17 (18) | 9 (9)
Cardiac arrest (Cardiac disorders) | 20 (20) | 20 (20)
Myocardial infarction (Vascular disorders) | 31 (34) | 26 (27)
Coronary Artery Disease (Vascular disorders) | 22 (25) | 22 (23)
Peripheral vascular disease (Vascular disorders) | 13 (15) | 15 (20)
Aortic stenosis (Cardiac disorders) | 2 (2) | 2 (2)
Mitral stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Mitral regurgitation (Cardiac disorders) | 5 (5) | 7 (8)
Tricuspid regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Valvular damage/Valvular insufficiency (Cardiac disorders) | 1 (1) | 4 (4)
Syncope (General disorders) | 17 (20) | 18 (25)
Dizziness (General disorders) | 4 (4) | 2 (2)
Chest pain - Ischemic (Vascular disorders) | 18 (18) | 18 (19)
Chest pain - Other (General disorders) | 28 (35) | 30 (34)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8)
Palpitations (Cardiac disorders) | 1 (1) | 1 (2)
Fatigue/Weakness (General disorders) | 0 (0) | 2 (2)
Multiple symptoms (General disorders) | 8 (8) | 16 (16)
Abdominal Aortic Aneurysm - Patient Condition - Cardiovascular (Cardiac disorders) | 3 (4) | 10 (12)
Amyloidosis - Patient Condition - Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Abdominal Aneurysm - Patient Condition - Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Sarcoidosis - Patient Condition - Cardiovascular (Cardiac disorders) | 1 (1) | 2 (2)
Internal Carotid Artery (ICA) - Patient Condition - Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Thoracic Aortic Aneurysm - Patient Condition - Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (TIA) (Vascular disorders) | 3 (3) | 3 (3)
Cerebrovascular Accident (CVA) - unspecifed (Vascular disorders) | 15 (15) | 20 (21)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 11 (11) | 4 (4)
Pulmonary Embolism (PE) (Vascular disorders) | 10 (10) | 7 (7)
Distal thromboemboli (Vascular disorders) | 0 (0) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Arterial/venous thrombolytic event (Vascular disorders) | 3 (3) | 1 (1)
Cerebrovascular Accident (CVA) - ischemic (Vascular disorders) | 6 (6) | 14 (15)
Cerebrovascular Accident (CVA) - hemorrhagic (Vascular disorders) | 3 (3) | 1 (1)
Pericardial effusion - Unrelated (non study) procedure or device (Cardiac disorders) | 1 (1) | 3 (3)
Pericarditis - Unrelated (non study) procedure or device (Cardiac disorders) | 0 (0) | 1 (1)
Hematoma - Unrelated (non study) procedure or device (Vascular disorders) | 3 (3) | 0 (0)
Hemorrhage - Unrelated (non study) procedure or device (Vascular disorders) | 0 (0) | 2 (2)
Pneumothorax - Unrelated (non study) procedure or device (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Infection - Unrelated (non study) procedure or device (Infections and infestations) | 2 (2) | 2 (2)
Pleural Effusion - Unrelated (non study) procedure or device (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Adverse reaction - General (General disorders) | 5 (5) | 3 (3)
Adverse reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Adverse reaction - Allergic reaction (General disorders) | 0 (0) | 1 (1)
Vasovagal reaction (General disorders) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 17 (22)
Adverse reaction - Medication (General disorders) | 1 (1) | 0 (0)
Alcohol Dependency - Patient Condition - Non-Cardiovascular (General disorders) | 1 (1) | 0 (0)
General Discomfort - Patient Condition - Non-Cardiovascular (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 32 (32) | 24 (24)
Systemic infection (Infections and infestations) | 46 (48) | 38 (46)
Fever and/or Virus (Infections and infestations) | 8 (8) | 8 (8)
Physical trauma (General disorders) | 11 (11) | 7 (8)
Abnormal laboratory values (General disorders) | 15 (17) | 15 (15)
Localized Infection (Infections and infestations) | 13 (15) | 9 (11)
Hematological (Blood and lymphatic system disorders) | 14 (15) | 23 (25)
Neurological (Nervous system disorders) | 19 (25) | 21 (27)
Gastrointestinal (Gastrointestinal disorders) | 82 (99) | 69 (102)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 94 (110) | 94 (113)
Abominal Pseudoanerysm with active extravasion - Whole Body (General disorders) | 0 (0) | 1 (1)
Obesity - Whole Body (General disorders) | 1 (1) | 0 (0)
PICC Line Malfunction - Whole Body (General disorders) | 0 (0) | 1 (1)
Sternal Wire Protrusion s/p CABG repair - Whole Body (General disorders) | 1 (1) | 0 (0)
Genitourinary (Renal and urinary disorders) | 18 (22) | 23 (28)
Renal (Renal and urinary disorders) | 34 (45) | 47 (52)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 44 (47) | 33 (42)
Psychological (Psychiatric disorders) | 7 (7) | 8 (8)
Integumentary (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (10)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 9 (12) | 8 (9)
Endocrine (Endocrine disorders) | 10 (11) | 15 (16)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (63) | 33 (37)
Multi-system failure (General disorders) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATP and Shock (N=1302) | Shock Only (N=1293)
Oversensing - RA PG System (Product Issues) | 2 (2) | 1 (1)
Undersensing - RA PG System (Product Issues) | 1 (1) | 0 (0)
Oversensing - RV PG System (Product Issues) | 1 (1) | 0 (0)
Impedance Out of Range - RV PG System (Product Issues) | 1 (1) | 0 (0)
Oversensing - Defibrillation - PG System (Product Issues) | 1 (1) | 0 (0)
Inappropriate Tachy Therapy - SVT - PG System Therapy (Product Issues) | 20 (25) | 40 (57)
Early ERI - Premature declaration - PG System Therapy (Product Issues) | 1 (1) | 0 (0)
Pacemaker Mediated Tachycardia - PG System Therapy (Product Issues) | 1 (1) | 4 (4)
Inadequate healing of incision site - PG System - Subject related (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psychological effect due to device therapy - PG System - Subject related (Psychiatric disorders) | 0 (0) | 1 (1)
Twiddler's Syndrome - PG System - Subject related (Psychiatric disorders) | 1 (1) | 0 (0)
Migration - PG System - Subject related (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Complex Regional Pain Syndrome and Frozen Shoulder - PG System - Patient Related (Product Issues) | 1 (1) | 0 (0)
Pain at Site - PG System - Patient Related (Product Issues) | 0 (0) | 1 (1)
Post-surgical wound discomfort/bruising/swelling (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Post-surgical infection (<=30 days post-implant) (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Thromboembolic events (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Oversensing - RA Lead (Product Issues) | 0 (0) | 2 (2)
Undersensing - RA Lead (Product Issues) | 0 (0) | 1 (1)
Unable to capture - RA Lead (Product Issues) | 1 (1) | 1 (1)
Elevated threshold - RA Lead (Product Issues) | 1 (1) | 0 (0)
Extracardiac stimulation - RA Lead (Product Issues) | 0 (0) | 1 (1)
Conductor coil fracture - RA Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Elevated threshold - RA Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Multiple signs - RA Lead (Product Issues) | 1 (1) | 0 (0)
Dislodgment - No reported signs - RA Lead (Product Issues) | 1 (1) | 1 (1)
Oversensing - RV Lead (Product Issues) | 0 (0) | 1 (1)
Elevated threshold - RV Lead (Product Issues) | 0 (0) | 1 (1)
Extracardiac stimulation - RV Lead (Product Issues) | 0 (0) | 1 (1)
Conductor coil fracture - RV Lead (Product Issues) | 1 (1) | 0 (0)
Insulation breach - RV Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Unable to capture - RV Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - Elevated threshold -RV Lead (Product Issues) | 1 (1) | 3 (4)
Dislodgment - Undersensing - RV Lead (Product Issues) | 0 (0) | 1 (1)
Dislodgment - No reported signs - RV Lead (Product Issues) | 2 (2) | 0 (0)
Impedance Out of Range - Defibrillation lead (Product Issues) | 1 (1) | 1 (1)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pericardial effusion - Procedure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Attempted coronary sinus lead placement - Lead - Procedure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
3rd degree AV block (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 4 (4)
Ventricular Fibrillation (VF) (Cardiac disorders) | 19 (23) | 28 (32)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 93 (150) | 117 (176)
Nonsustained Ventricular Tachycardia (NSVT) (Cardiac disorders) | 153 (178) | 150 (178)
Atrial Fibrillation (AF) (Cardiac disorders) | 100 (110) | 96 (120)
Atrial Flutter (Cardiac disorders) | 9 (10) | 9 (9)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 2 (2)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 67 (93) | 53 (92)
Junctional ectopic rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 2 (2) | 3 (3)
Arrhythmia Not Specified - Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Intraventricular Conduction Disorder - Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Prolonged Q-T Interval - Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia patient reported - Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
VF with Syncope - Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
VT with Syncope - Arrhythmia (Cardiac disorders) | 7 (8) | 10 (11)
Dizziness - Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain - Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Dyspnea - Heart failure (Cardiac disorders) | 6 (6) | 11 (13)
Peripheral edema - Heart failure (Cardiac disorders) | 2 (2) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Renal insufficiency/failure - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 6 (6) | 9 (10)
Multiple heart failure symptoms (Cardiac disorders) | 13 (13) | 16 (16)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 8 (8) | 6 (6)
Hypertension/Hypertensive Crisis (Vascular disorders) | 1 (1) | 2 (2)
Myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 20 (21) | 17 (18)
Dizziness (General disorders) | 10 (11) | 15 (16)
Chest pain - Ischemic (Vascular disorders) | 1 (1) | 1 (1)
Chest pain - Other (General disorders) | 7 (7) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Multiple symptoms (General disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (TIA) (Vascular disorders) | 2 (2) | 0 (0)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Arterial/venous thrombolytic event (Vascular disorders) | 1 (1) | 0 (0)
Pericarditis - Unrelated (non study) procedure or device (Cardiac disorders) | 0 (0) | 1 (1)
Hematoma - Unrelated (non study) procedure or device (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage - Unrelated (non study) procedure or device (Vascular disorders) | 1 (1) | 0 (0)
Infection - Unrelated (non study) procedure or device (Infections and infestations) | 1 (1) | 0 (0)
Puncture Site Ulcer - Unrelated Procedure/Device (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Adverse reaction - General (General disorders) | 1 (1) | 0 (0)
Adverse reaction - Hypotension (Vascular disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Adverse reaction - Medication (General disorders) | 1 (1) | 0 (0)
Abdominal Pain - Patient Condition - Non-Cardiovascular (General disorders) | 1 (1) | 0 (0)
Dehydration - Patient Condition - Non-Cardiovascular (General disorders) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1) | 2 (2)
Fever and/or Virus (Infections and infestations) | 0 (0) | 1 (1)
Physical trauma (General disorders) | 3 (3) | 1 (1)
Abnormal laboratory values (General disorders) | 3 (5) | 3 (4)
Localized Infection (Infections and infestations) | 0 (0) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Neurological (Nervous system disorders) | 4 (4) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 4 (5) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Genitourinary (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal (Renal and urinary disorders) | 3 (3) | 3 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Psychological (Psychiatric disorders) | 0 (0) | 1 (2)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 3 (3) | 2 (2)
Endocrine (Endocrine disorders) | 3 (3) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
COVID-19 led to an increase in missed visits, late visits, withdrawals and several site personnel changes.

Additional ATP programming options were not evaluated, only the effect of a single ATP burst of 8 pulses at 88% cycle length.

The differential delay to shock between arms due to ATP (~3 seconds) may have led to more shocks in the Shock Only arm.

The utility of ATP in other primary prevention indications was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Sponsor may extend the review period for another 90 days to take steps to protect its intellectual property interests, or to remove any language detrimental to Sponsor's intellectual property interests.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02923726/Prot_SAP_000.pdf